CLINICAL TRIAL: NCT06186596
Title: Patient Self-Administered Intralesional Injections of Triamcinolone for Acne Vulgaris
Brief Title: Self-Administered Intralesional Injections for Acne
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ACOM Labs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATM-2301
Record Dates: First submitted 2023-12-05; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention (Experimental): All subjects will receive standard-of-care intralesional injection with triamcinolone using an Injection Assistance Device (i.e., for self-administered intralesional injections) at Visit 1 (Day 1). Subjects will then submit photos via secure photographic app for asynchronous follow up on Day 2 (24-hours post-injection), Day 3 (48-hours post-injection), Day 4 (72-hours post-injection), Day 7, and Day 14.
  Interventions: Device: Triamcinolone delivered via injection assistance device

INTERVENTIONS:
Device: Triamcinolone delivered via injection assistance device — 0.1mL of 1% to 2% triamcinolone solution will be delivered to up to 3 facial inflammatory acne lesions

SUMMARY:
The goal of this clinical trial is to test the safety of intralesional injections of triamcinolone self-administered into acne lesions via an injection assistance device. The main question[s] it aims to answer are:

* is use of the injection assistance device safe?
* is delivery of triamcinolone to acne lesions via the injection assistance device efficacious?

Participants will self-inject low dose triamcinolone into acne lesions and track lesion response via photos and survey for 14 days following injection.

DETAILED DESCRIPTION:
This is an open-label, prospective, single-arm study. Approximately 150 subjects will be enrolled at approximately 3 study sites.

All subjects will receive standard-of-care intralesional injection with triamcinolone using an Injection Assistance Device (i.e., for self-administered intralesional injections) at Visit 1 (Day 1). Subjects will then submit photos via secure photographic app for asynchronous follow up on Day 2 (24-hours post-injection), Day 3 (48-hours post-injection), Day 4 (72-hours post-injection), Day 7, and Day 14.

Efficacy assessments (target lesion assessments) will be conducted remotely by the Investigator at time of each photo submission. Subjects will conduct lesion pain assessments and satisfaction assessments at the time of each remote check-in. Participants will be invited to also have additional photography captured by the study team at the study site or at a location as per participants' convenience.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient, male or female of any race, 18 years of age or older. Female subjects of childbearing potential must have a negative UPT at Baseline.
2. Diagnosed with facial acne vulgaris.
3. At least one (1) identifiable inflammatory lesion that, in the opinion of the investigator, is clinically indicated for standard-of-care intralesional injection(s) of triamcinolone.
4. Owner of smartphone with capacity for front-facing photography and app download from Apple App Store or Google Play.
5. Able to follow study instructions and likely to comply with virtual follow-up requirements.
6. In good general health as determined by medical history at the time of screening (Investigator discretion).
7. Sign the IRB-approved ICF (including HIPAA authorization) prior to any study-related procedures being performed.

Exclusion Criteria:

1. Female subjects who are pregnant or breast-feeding.
2. Known hypersensitivity or previous allergic reaction to any constituent of triamcinolone injection.
3. Active cutaneous viral infection in any treatment area at Baseline.
4. Have concomitant skin disease or infection (other than acne) or presence of skin comorbidities in the areas of skin where study device will be used.
5. History of poor cooperation or unreliability (Investigator discretion).
6. Subjects who are investigational site staff members or family members of such employees.
7. Exposure to any other investigational device within 30 days prior to Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events following device use | 14 days
  Adverse events associated with device use for 14 days following injection

SECONDARY OUTCOMES:
Target Lesion Pain | 14 days
  For each inflammatory lesion injected, lesion pain will be assessed by the subject 0 to 10 scale, where 0 is no pain and 10 is worst imaginable pain. Lesion pain at Baseline will be recorded prior to injection(s). The occurrence of inflammatory lesion pain is expected and will not be considered an AE.
Target Lesion Injection Pain | baseline and 5 min following injection
  Injection Site Pain during injection will be assessed immediately after the injection of the first target lesion and at 5 minutes post-injection. The occurrence of injection site pain is expected and will not be considered an AE. For each inflammatory lesion injected, lesion pain will be assessed by the subject 0 to 10 scale, where 0 is no pain and 10 is worst imaginable pain.
Target Lesion Change (subject) | 24 hours - 14 days
  The subject will assess subjective improvement seen with each target lesion compared to Baseline.
  1. Clear (100%)
  2. Almost clear (90% to <100%)
  3. Marked improvement (75% to <90%)
  4. Moderate improvement (50% to <75%)
  5. Fair improvement (25% to <50%)
  6. No change
  7. Worse
Subject satisfaction or dissatisfaction with treatment assessed via a 5-grade scale | 24 hours - 14 days
  Satisfaction or dissatisfaction with will be assessed by the subject using the following subjective 5-grade scale as detailed below. Subject will be instructed: "Rate your level of satisfaction with the effect of study treatment on inflammatory acne lesions by using the following scale":
  1. Very satisfied
  2. Satisfied
  3. Neither satisfied nor dissatisfied
  4. Dissatisfied
  5. Very dissatisfied
Target Lesion Erythema | baseline - 14 days
  Investigator will assess severity of erythema for each target lesion on a 0 (no erythema) to 4 (very severe erythema) scale.
  0: No Erythema
  1. Mild Erythema
  2. Moderate Erythema
  3. Severe Erythema
  4. Very Severe Erythema
Target Lesion Severity | baseline - 14 days
  Investigator will assess severity of each target lesion on a 0 (none) to 4 (very severe) scale.
  0: None
  1. Mild
  2. Moderate
  3. Severe
  4. Very Severe
Target Lesion Change | 24 hours - 14 days
  Investigator will assess improvement of each target lesion on a 1 (100% clear) to 7 (worse) scale.
  1. Clear (100%)
  2. Almost clear (90% to <100%)
  3. Marked improvement (75% to <90%)
  4. Moderate improvement (50% to <75%)
  5. Fair improvement (25% to <50%)
  6. No change
  7. Worse

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Center For Dermatology Clinical Research, Inc, Fremont, California
  - Skin Care Research, Boca Raton, Florida
  - Skin Care Research, Hollywood, Florida

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/96/NCT06186596/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/96/NCT06186596/ICF_001.pdf